CLINICAL TRIAL: NCT02946242
Title: Development Of Medical Ultrasound Systems, Accessories, And Components - GE Bangalore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110.08-2015-GES-0004
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2022-07

CONDITIONS: Ultrasound Exams

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- General Ultrasound Exam (Other): Each subject may elect to participate in up to five (5) study scans per day lasting up to 60 cumulative minutes each with approximately a 15 minute break before starting another study scan. Ophthalmic scanning will be limited to no more than 15 cumulative minutes of scan time per eye, per day.
  Interventions: Device: Ultrasound Exam

INTERVENTIONS:
Device: Ultrasound Exam — Subjects will be scheduled to attend up to up to five (5) ultrasound scans per day lasting up to 60 cumulative minutes each with approximately a 15 minute break before starting another study scan (limited to 15 cumulative minutes of scan time per eye, per day for ophthalmic scanning) as long as they remain eligible per the study inclusion and eligibility criteria.

SUMMARY:
Ultrasound devices components and accessories are under continuous development in order to optimize, validate and improve the devices, including improving the quality of images. In this study, GEHC proposes to collect data in order to achieve the following

1. Aim 1: Perform iterative evaluations of the device (including features, accessories and components) to optimize device performance, assess feasibility of new features, and to perform testing necessary to support product and technology development;
2. Aim 2: Perform activities to support design validation and/or to confirm user requirements and specifications have been met, as per design controls and other applicable requirements;
3. Aim 3: Evaluate device complaints and analyze potential causes. There is no animal or phantom model that is adequate to accomplish these aims; therefore human subjects are required.

Due to the inherently varied nature of study data, specific data points will be recorded on a per-case basis and the study final report will summarize at minimum number and type of study scans conducted. Electronic image data may be collected. The number and type of safety issues, including adverse events (AEs) and serious adverse events (SAEs) will be reported. Unexpected device issues that occur outside of expected and controlled engineering optimization will be reported.

DETAILED DESCRIPTION:
Subjects will be considered enrolled that provide written informed consent to participate, and with thereafter be scheduled to attend up to up to five (5) ultrasound scans per day lasting up to 60 cumulative minutes each with approximately a 15 minute break before starting another study scan (limited to 15 cumulative minutes of scan time per eye, per day for ophthalmic scanning) as long as they remain eligible per the study inclusion and eligibility criteria. Vital sign information about subjects may be collected and subjects will be positioned for scanning of a variety of target anatomic areas using a variety of non-invasive, transcutaneous techniques, such as scanning abdominal, musculoskeletal, breast(s), peripleural, transcranial, cervical/neck, cardiac, ophthalmic, vascular, extremity, soft tissue, and other accessible anatomical regions. The subject will be monitored for adverse events throughout the research study scan. The resultant images and associated data will be recorded and stored as part of study data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Able and willing to provide written informed consent in accordance with the PNDT Act in India
3. Able to understand and respond in English
4. General Electric (GE) employee or contractor at the John F. Welch Technology Centre (JFWTC) facility.

Exclusion Criteria:

1. Direct employee or contractor of the General Electric (GE) Ultrasound business at the John F. Welch Technology Centre (JFWTC) facility
2. If female, pregnant or unsure of her pregnancy status per self-report.
3. Is not able to or would be put at additional risk from completing study activities, in the opinion of the study staff.
4. Subjects who have an electronic medical device at the time of the study scan (such as pacemaker, implantable cardioverter/defibrillator, insulin pump, cochlear implant, or other implanted electronic medical device).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Completion of diagnostic ultrasound exam | 1 day
  Parameters, features, and operator notes from the exam will be recorded to support diagnostic exam completion

OTHER OUTCOMES:
Exam completion data may be stratified by exam type/indication based on actual site accrual. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Gupta, MD, Principal Investigator — GE Healthcare
Locations (1):
- Wipro GE Healthcare Pvt. Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02946242/Prot_000.pdf